CLINICAL TRIAL: NCT06350838
Title: A Phase I Clinical Study to Investigate the Safety and Tolerance of Therapeutic Bacillus Calmette-Guerin( BCG) in Postoperative Adjuvant Therapy in Subjects With Moderate to High-risk Non-muscular Invasive Bladder Cancer (NMIBC)
Brief Title: Clinical Study to Investigate the Safety and Tolerance of Therapeutic BCG in Postoperative Adjuvant Therapy in Subjects With Moderate to High-risk Non-muscular Invasive Bladder Cancer (NMIBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu CoenBiotech Co., Ltd (Industry)
Collaborators: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN-BCG-I
Record Dates: First submitted 2024-01-28; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Non-muscular Invasive Bladder Cancer
Keywords: Non-muscular invasive bladder cancer; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Therapeutic Uses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medium/high-risk non-muscle invasive bladder cancer (NMIBC) (Experimental): Medium/high-risk NMIBC (Ta, T1 or Tis) suitable for intravesical BCG treatment.Three phases included: screening period (28 days before the first dose), observation period (6 weeks) and safety follow-up period (7 days after the last dose).
  Interventions: Drug: BCG for Therapeutic Use

INTERVENTIONS:
Drug: BCG for Therapeutic Use — Take 120 mg BCG for treatment, dissolved in 40 ~ 50 mL normal saline, bladder perfusion through catheter. The injection was performed once a week for 6 consecutive times.
  Other Names: BCG

SUMMARY:
Phase I clinical study to investigate the safety and tolerance of therapeutic BCG in postoperative adjuvant therapy in subjects with moderate to high-risk non-muscular invasive bladder cancer (NMIBC)

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety and tolerance, pharmacokinetic characteristics, ablative status, and immune response characteristics of the therapeutic BCG in postoperative adjuvant therapy in subjects with moderate and high-risk non-invasive bladder cancer (NMIBC).

The study consisted of three phases: screening period, administration observation period and safety follow-up period. subjects will be treated with 120 mg BCG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were ≥18 years old and ≤85 years old, male or female;
* Subjects with non-myoinvasive bladder uroepithelial carcinoma initially diagnosed by histology [T1, Ta, or Tis stage (carcinoma in situ)] and assessed as moderate to high-risk non-myoinvasive bladder uroepithelial carcinoma requiring BCG injection adjuvant therapy according to the Guidelines for Bladder Cancer Diagnosis and Treatment (2022 edition); (Subjects considered for secondary resection may be included in the study after completion of secondary resection and pathology results confirm moderate or high risk non-myoinvasive bladder cancer);
* ECOG score: 0-2;
* Clinical laboratory tests meet the following characteristics:

  1. Blood routine: no hematopoietic growth factor or transfusion support was used within 14 days prior to enrollment, including: absolute neutrophil value (ANC) ≥1500/mm3 or ≥1.5×109/L; Platelets ≥100000/mm3 or 100×109/L; Hemoglobin ≥9 g/dL.
  2. Liver function: total serum bilirubin ≤1.5× upper limit of normal range (ULN), total serum bilirubin <3×ULN in subjects with Gilbert syndrome, aspartate and alanine aminotransferase (AST and ALT) ≤2.5×ULN.
  3. Renal function: defined as creatinine clearance ≥45 to 50 mL/min as estimated by the Cockcroft Gault formula.
  4. Coagulation function: Activated partial thromboplastin time (APTT) ≤1.5×ULN, International Normalized ratio (INR) ≤1.5×ULN
* The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Any of the following:

  1. Patients who are using immunosuppressive drugs, hormone drugs, or radiation therapy that the investigator has determined to be likely to cause systemic BCG disease reactions (patients who hormone injections for thyroid/adrenal resection may be included);
  2. Allergic to BCG vaccine or BCG products;
  3. Have active TB changes or are receiving anti-TB therapy;
  4. Known or suspected intraoperative perforation of the bladder; e Serious gross hematuria before administration was judged by the investigator, and the surgical wound was suspected to have not healed.

  f. The evaluators were judged to be associated with cystitis, or had previously received other bladder perfusion drugs, and were expected to have severe bladder irritation.

  f. Patients with a history of severe adverse reactions to BCG (BCG) sepsis or systemic infection; g. Complete bladder incontinence, defined as the use of six or more pads in a 24-hour period; h. Complete bladder incontinence, defined as the use of six or more pads in a 24-hour period;
* Combined with other genitourinary tumors or malignancies of other organs;
* Accompanied by serious diseases of cardiovascular and cerebrovascular, lung, liver, kidney and other important organs, or severe hypertension or diabetes that researchers judge can not be controlled clinically;
* Patients suffering from acute infectious diseases at the time of screening;
* Evidence of Myoinvasive locally advanced or metastatic urothelial carcinoma, or extrinsic non-Myoinvasive urothelial metastasized cell carcinoma, as determined by the investigator;
* Study participants who had received chemotherapy, radiation therapy, or anti-tumor immunotherapy within 4 weeks prior to treatment (except for immediate postoperative bladder infusion chemotherapy);
* Pregnant or lactating women;
* Subjects who are unable to use effective contraception during the trial period and within 3 months after the last dose;
* Participants who had participated in clinical trials of other therapeutic drugs within 1 month prior to enrollment;
* Known opioid or alcohol dependence;
* Human immunodeficiency virus (HIV) antibody, syphilis specific antibody positive, acute or chronic active hepatitis B (hepatitis B surface antigen (HBsAg) positive, and peripheral blood hepatitis B copy number ≥103/mL), hepatitis C virus (HCV) antibody positive (HCV copy number ≥10/mL);
* Patients with mental disorders or poor compliance as judged by the investigator;
* Any conditions that the investigator believes may increase risk to the subject or interfere with the execution of the clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events(TEAE) and serious Treatment-Emergent Adverse Events; | 6 weeks
  Probability of AE and SAE after administration.
Effects on clinical laboratory tests index of blood biochemistry, such as the concentration of alanine aminotransferase (ALT). | 6 weeks
  Probability of abnormal laboratory parameters of blood biochemistry compared with baseline，such as the concentration of alanine aminotransferase (ALT).
Effects on clinical laboratory tests index of blood routine, such as white blood cell count, red blood cell count, platelet count. | 6 weeks
  Probability of abnormal laboratory parameters of blood routine compared with baseline, such as white blood cell count, red blood cell count, platelet count.
Effects on clinical laboratory tests index of coagulation function, such as activated partial thromboplastin time (APTT). | 6 weeks
  Probability of abnormal laboratory parameters of coagulation function compared with baseline，such as activated partial thromboplastin time (APTT).
Effects on clinical laboratory tests index of urine routine, such as white urine albumin count, urine red blood cell count. | 6 weeks
  Probability of abnormal laboratory parameters of urine routine compared with baseline，such as urine albumin count, urine red blood cell count.
Effects on vital signs,such as temperature. | 6 weeks
  Probability of abnormal laboratory parameters of vital signs compared with baseline，such as temperature(℃).
Effects on P wave, QRS complex, QT interval and so on by 12-lead electrocardiogram. | 6 weeks
  Probability of abnormal laboratory parameters compared with baseline， including P wave, QRS complex, QT interval and so on by 12-lead electrocardiogram.
Effects on the periodic activity of echocardiography，such as the heart wall recorded as the relationship curve between the corresponding activity and time of each structure. | 6 weeks
  Probability of abnormal laboratory parameters of echocardiography compared with baseline，such as the heart wall recorded as the relationship curve between the corresponding activity and time of each structure.
Effects on physical examination, refers to the detection and measurement of the development level of human form, structure and function. | 6 weeks
  Probability of abnormal laboratory parameters of examination compared with baseline，such as any abnormalities in the skin.

SECONDARY OUTCOMES:
Exposure condition of the test drug in the blood, refer to plasma concentration of the test drug(BCG). | 6 weeks
  Exposure to the test drug in the blood，detecting the amount and concentration of drug.
Shedding condition of the test drug in urine. | 6 weeks
  Exposure to the test drug and in urine，detecting the amount and concentration of drug.
To investigate the immune response characteristics of therapeutic BCG in patients with moderate and high- risk non-invasive bladder cancer after surgery. | 6 weeks
  The amount and concentration levels of IL-2, IL-6, IL-8, IL-12, IFN-γ, and TNF in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided